CLINICAL TRIAL: NCT06426719
Title: Efficiency of Using Osseodensification Protocol for Alveolar Ridge Expansion in Edentulous Alveolar Ridges
Brief Title: Efficiency of Using Osseodensification Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Magdy Mostafa Shehata (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Mohamed Magdy Mostafa Shehata, doctor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 28908210103756
Record Dates: First submitted 2024-05-09; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Alveolar Bone Resorption
Keywords: Densah burs; Osseodensification; OsseoHand Osteotomes; alveolar ridge wideninig

STUDY DESIGN:
Intervention Model Description: a new technique used to provide sufficient alveolar ridge width and enhance bone quality at horizontally deficient maxillary alveolar ridges prior to implant placement. the new technique uses specially designed burs called Densah burs that act by causeing bone compaction rather than bone removing from the osteotomy site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group osseodensification (Experimental): the group in which alveloalr ridge widening is done using densah burs, it is the study group
  Interventions: Procedure: Alveolar ridge wideninig via applying osseodensification protocol using densah burs
- conventional osteotome group (Active Comparator): the group in which alveolar ridge expansion is done using hand driven osteotomes . it is the conventional froup
  Interventions: Procedure: Alveolar ridge widening via hand osteotomes

INTERVENTIONS:
Procedure: Alveolar ridge wideninig via applying osseodensification protocol using densah burs — alveolar ridge expansion using densah burs in horizontally deficient maxillary alveolar ridges prior to dental implants insertion
  Arms: intervention group osseodensification
Procedure: Alveolar ridge widening via hand osteotomes — Alveolar ridge expansion using hand driven osteotomes in horizontally deficient maxillary alveolar ridges prior to dental Implant insertion
  Arms: conventional osteotome group

SUMMARY:
the goal of this clinical trial is to learn if the new osseo-densification technique works to provide enough bone width and quality prior to implant placement in the upper jaw the main question it aims to answer is: Is the use of osseo-densification protocol better than the standard alveolar ridge widening techniques; regarding efficiency and comfort in obtaining sufficient alveolar ridge width in horizontally atrophic alveolar ridges?

DETAILED DESCRIPTION:
a new osseo-densification protocol using specially designed Densah burs was compared to conventional hand Osteotome technique to test its efficiency in providing sufficient bone quantity and quality in cases of horizontally deficient maxillary edentulous alveolar ridge sites that require expansion prior to dental implant placement

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* In cases of an initial ridge width ≤ 5mm that contains ≤ 2mm of trabecular bone core.
* Alveolar ridges with narrow crest and wider base.

Exclusion Criteria:

* Uncontrolled diabetic patients
* Heavy Smokers
* Patients suffering from osteoporosis
* Patients receiving chemo or radio therapy
* Patients suffering from bleeding disorders
* Patients suffering from intraosseous lesions at the proposed site of implant
* Patients with insufficient alveolar bone hight less than 10 mm.
* Resorbed ridge with a narrow base.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
efficiency of ridge widening technique | intraoperative and within 3 days post operative
  the amount of ridge width gain is measured both clinically via a caliber and radiographically on CBCT

SECONDARY OUTCOMES:
primary stability of implant | intra-operative after dental implant placement
  the primary stability of the inserted dental implant is measured via osstell device
length of surgical procedure | During surgery
  the time required for completion of the surgical procedure is measured in minutes using stop watch
Value of pain | Immediate post operative
  the degree of pain or discomfort examined by the patient during the ridge widening procedure is recorded using a visual scale where 0 represents no pain while 1 minimum pain and 10 is maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Shehata, Principal Investigator — Cairo University
Locations (1):
- Mohamed Magdy Mostafa shehata, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: within 6 months from publication
Access Criteria: IDP will be shared with researchers and clinical investigators who require them for further systematic review or retrograde studies via contacting the principal investigator through email

REFERENCES:
- [Result] Tian JH, Neiva R, Coelho PG, Witek L, Tovar NM, Lo IC, Gil LF, Torroni A. Alveolar Ridge Expansion: Comparison of Osseodensification and Conventional Osteotome Techniques. J Craniofac Surg. 2019 Mar/Apr;30(2):607-610. doi: 10.1097/SCS.0000000000004956. PMID 30507887
- [Result] Bassetti MA, Bassetti RG, Bosshardt DD. The alveolar ridge splitting/expansion technique: a systematic review. Clin Oral Implants Res. 2016 Mar;27(3):310-24. doi: 10.1111/clr.12537. Epub 2015 Jan 14. PMID 25586966
- [Result] Jha N, Choi EH, Kaushik NK, Ryu JJ. Types of devices used in ridge split procedure for alveolar bone expansion: A systematic review. PLoS One. 2017 Jul 21;12(7):e0180342. doi: 10.1371/journal.pone.0180342. eCollection 2017. PMID 28732054
- [Result] Inchingolo AD, Inchingolo AM, Bordea IR, Xhajanka E, Romeo DM, Romeo M, Zappone CMF, Malcangi G, Scarano A, Lorusso F, Isacco CG, Marinelli G, Contaldo M, Ballini A, Inchingolo F, Dipalma G. The Effectiveness of Osseodensification Drilling Protocol for Implant Site Osteotomy: A Systematic Review of the Literature and Meta-Analysis. Materials (Basel). 2021 Feb 28;14(5):1147. doi: 10.3390/ma14051147. PMID 33671038
- [Result] Padhye NM, Padhye AM, Bhatavadekar NB. Osseodensification -- A systematic review and qualitative analysis of published literature. J Oral Biol Craniofac Res. 2020 Jan-Mar;10(1):375-380. doi: 10.1016/j.jobcr.2019.10.002. Epub 2019 Nov 2. PMID 31737477
- [Result] Witek L, Alifarag AM, Tovar N, Lopez CD, Gil LF, Gorbonosov M, Hannan K, Neiva R, Coelho PG. Osteogenic parameters surrounding trabecular tantalum metal implants in osteotomies prepared via osseodensification drilling. Med Oral Patol Oral Cir Bucal. 2019 Nov 1;24(6):e764-e769. doi: 10.4317/medoral.23108. PMID 31655837
- [Result] Starch-Jensen T, Becktor JP. Maxillary Alveolar Ridge Expansion with Split-Crest Technique Compared with Lateral Ridge Augmentation with Autogenous Bone Block Graft: a Systematic Review. J Oral Maxillofac Res. 2019 Dec 30;10(4):e2. doi: 10.5037/jomr.2019.10402. eCollection 2019 Oct-Dec. PMID 32158526
- [Result] Demetriades N, Park JI, Laskarides C. Alternative bone expansion technique for implant placement in atrophic edentulous maxilla and mandible. J Oral Implantol. 2011 Aug;37(4):463-71. doi: 10.1563/AAID-JOI-D-10-00028. Epub 2010 Jul 21. PMID 20662673